CLINICAL TRIAL: NCT01691768
Title: Open-Label Randomized Controlled Trial to Assess the Implementation Effectiveness and Safety of 1% Tenofovir Gel Provision Through Family Planning Services in KwaZulu-Natal, South Africa
Brief Title: Implementation Effectiveness and Safety of Tenofovir Gel Provision Through Family Planning Services
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: CONRAD (Other); Gilead Sciences (Industry); FHI 360 (Other); Institute for Healthcare Improvement (Other)
Responsible Party: Principal Investigator, Dr Quarraisha Abdool Karim, Associate Scientific Director, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAPRISA008; NCT01645813 (obsolete NCT alias)
Record Dates: First submitted 2012-07-05; First posted 2012-09-25 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: HIV
Keywords: microbicides; women; HIV prevention; PrEP; Tenofovir gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): 1% tenofovir gel provision through a public sector family planning services with 2-3 monthly provision and monitoring and the use of Quality Improvement methodology to promote reliable service delivery
  Interventions: Drug: 1% tenofovir gel
- Control (Active Comparator): monthly 1% tenofovir gel provision and monitoring through CAPRISA research clinics
  Interventions: Drug: 1% tenofovir gel

INTERVENTIONS:
Drug: 1% tenofovir gel — Participants will be randomized to receive 1% tenofovir gel through either:
  * Public sector family planning services with 2-3 monthly provision and monitoring of 1% tenofovir gel and the use of QI methodology to promote reliable service delivery (intervention arm), or
  * The CAPRISA research clinics with monthly provision and monitoring of 1% tenofovir gel (control arm).

SUMMARY:
The purpose of this study is to assess the effectiveness of an implementation model which integrates tenofovir gel provision into existing family planning services.

DETAILED DESCRIPTION:
The CAPRISA 008 trial is a two-arm, open-label, randomized controlled trial that is being conducted at the CAPRISA eThekwini and CAPRISA Vulindlela Clinics and their neighboring public sector family planning services in KwaZulu-Natal, South Africa. Up to 700 consenting sexually active, HIV-uninfected women aged 18 years and older who previously participated in an antiretroviral (ARV) prevention study will be enrolled and followed for a maximum 30 months. All women will be provided with 1% tenofovir gel but will be randomised to either receive their gel through a public sector family planning services with 2-3 monthly provision (intervention arm) or through the CAPRISA research clinics with monthly provision (control arm).

All women in the trial will be provided with the standard package of HIV prevention and reproductive health services. Participants in both study arms will be provided with a supply of single-use, pre-filled applicators of 1% tenofovir gel. While in the study, participants will be advised and supported to follow the CAPRISA 004 pre- and post-dosing strategy, namely BAT24, where the first dose of tenofovir gel is applied within 12 hours before anticipated coitus and a second dose as soon as possible but within 12 hours after coitus, with a maximum of two doses of gel in a 24-hour period.

The primary objective of this trial is to assess the effectiveness of an implementation model for tenofovir gel provision through family planning services.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Women who previously participated in an ARV prevention study
* Currently utilizing or agreeing to attend designated public sector family planning services
* Able and willing to provide first person informed consent to be screened for, and to enroll in, the study
* Able and willing to provide adequate locator information for study retention purposes
* Sexually active (at least one coital act in the last 3 months prior to screening)
* HIV negative (by HIV testing performed by study staff within 30 days of enrollment)
* Negative pregnancy test performed by study staff within 21 days of enrollment
* Agree to use a non-barrier form of contraceptive
* Agree to adhere to study visits and procedures

Exclusion Criteria:

* Has a creatinine clearance < 50ml/min
* Has any other condition that, based on the opinion of the Investigator or designee, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quarraisha Abdool Karim, PhD, Principal Investigator — Centre for the AIDS Programme of Research in South Africa
Locations (2):
- South Africa (2):
  - CAPRISA eThekwini Clinical Research Site, Durban, KwaZulu-Natal
  - CAPRISA Vulindlela Clinical Research Site, Pietermaritzburg, KwaZulu-Natal

REFERENCES:
- [Background] Abdool Karim Q, Abdool Karim SS, Frohlich JA, Grobler AC, Baxter C, Mansoor LE, Kharsany AB, Sibeko S, Mlisana KP, Omar Z, Gengiah TN, Maarschalk S, Arulappan N, Mlotshwa M, Morris L, Taylor D; CAPRISA 004 Trial Group. Effectiveness and safety of tenofovir gel, an antiretroviral microbicide, for the prevention of HIV infection in women. Science. 2010 Sep 3;329(5996):1168-74. doi: 10.1126/science.1193748. Epub 2010 Jul 19. PMID 20643915
- [Derived] Mngadi KT, Singh JA, Mansoor LE, Wassenaar DR. Undue inducement: a case study in CAPRISA 008. J Med Ethics. 2017 Dec;43(12):824-828. doi: 10.1136/medethics-2016-103414. Epub 2017 Mar 27. PMID 28348164
- [Derived] Mansoor LE, Abdool Karim Q, Mngadi KT, Dlamini S, Montague C, Nkomonde N, Mvandaba N, Baxter C, Gengiah TN, Samsunder N, Dawood H, Grobler A, Frohlich JA, Abdool Karim SS. Assessing the implementation effectiveness and safety of 1% tenofovir gel provision through family planning services in KwaZulu-Natal, South Africa: study protocol for an open-label randomized controlled trial. Trials. 2014 Dec 19;15:496. doi: 10.1186/1745-6215-15-496. PMID 25527071
- See also: Centre for the AIDS Programme of Research in South Africa web site — http://www.caprisa.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 448 were assessed for eligibility and 382 were randomized. However, only 372 were eligible for study participation. Of the 10 who were ineligibly enrolled: 6 were HIV positive at enrollment, 2 were co-enrolled in another trial, 1 had no post-randomization follow-up data and 1 was pregnant at enrollment.
Groups:
- Intervention: 1% tenofovir gel provision through a public sector family planning services with 2-3 monthly provision and monitoring and the use of Quality Improvement methodology to promote reliable service delivery
  1% tenofovir gel: Participants will be randomized to receive 1% tenofovir gel through either:
  * Public sector family planning services with 2-3 monthly provision and monitoring of 1% tenofovir gel and the use of QI methodology to promote reliable service delivery (intervention arm), or
  * The CAPRISA research clinics with monthly provision and monitoring of 1% tenofovir gel (control arm).
- Control: monthly 1% tenofovir gel provision and monitoring through CAPRISA research clinics
  1% tenofovir gel: Participants will be randomized to receive 1% tenofovir gel through either:
  * Public sector family planning services with 2-3 monthly provision and monitoring of 1% tenofovir gel and the use of QI methodology to promote reliable service delivery (intervention arm), or
  * The CAPRISA research clinics with monthly provision and monitoring of 1% tenofovir gel (control arm).
Period: Overall Study
Arm/Group | Intervention | Control
Started | 189 | 183
Completed | 174 | 167
Not Completed | 15 | 16
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Relocated | 0 | 1
Not completed — Investigator decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat population was analyzed. All participants who were randomized and met the pre-enrollment eligibility criteria.
Groups:
- Intervention: 1% tenofovir gel provision through a public sector family planning services with 2-3 monthly provision and monitoring and the use of QI methodology to promote reliable service delivery
  1% tenofovir gel: Participants will be randomized to receive 1% tenofovir gel through either:
  * Public sector family planning services with 2-3 monthly provision and monitoring of 1% tenofovir gel and the use of QI methodology to promote reliable service delivery (intervention arm), or
  * The CAPRISA research clinics with monthly provision and monitoring of 1% tenofovir gel (control arm).
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 189 | 183 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5.8) | 29.3 (5.3) | 29.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 183 | 372
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 189 | 183 | 372
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 189 | 183 | 372
Sex acts in past 30 days [Median (Inter-Quartile Range); unit: Acts] | 4 [3 to 8] | 4 [2 to 8] | 4 [2 to 8]
Contraception [Count of Participants; unit: Participants]
  Injectable | 139 | 140 | 279
  Oral | 43 | 32 | 75
  Sterilized | 7 | 11 | 18
HSV-2 prevalence [Count of Participants; unit: Participants] — Population: A total of 9 participants had equivocal results and 2 had missing results.
  Participants
    number analyzed (Participants) | 182 | 179 | 361
    (all) | 174 | 159 | 333
HPV prevalence [Count of Participants; unit: Participants] — Population: Total of 5 participants had equivocal and 2 had missing results.
  Participants
    number analyzed (Participants) | 186 | 179 | 365
    (all) | 20 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Returned Used Applicators Per Month (i.e in 30 Days)
Description: The primary endpoint is the mean number of returned used applicators per month. Since participants in the intervention arm followed two and three monthly schedule (as opposed to monthly in the intervention arm), the number of returned used applicators per month for each participant will be estimated as the total number of returned applicators at that visit divided by the number of days since the previous visit, multiplied by 30. Thus a uniform distribution of gel use will be assumed in participants whom we did not see monthly. Intent to treat and per protocol analyses were carried out of this outcome. Intent to treat population includes all participants who were randomized, met pre-randomization eligibility criteria and who have post-enrollment follow-up data. The per protocol population is a subset of the intent to treat population.The per-protocol analysis excluded visits where no gel had been dispensed for >120 days.
Time Frame: Between 2012 to 2015, up to 28 months
Population: Intent to treat population and the per protocol population (excluding all subsequent data collected from participants who were not dispensed product for more than 120 days).
Measure: Least Squares Mean (95% Confidence Interval); unit: Used gel applicators per month
Arm/Group | Intervention | Control
Number analyzed (Participants) | 189 | 183
Used gel applicators per month
  Intent to treat analyses | 5.2 [4.7 to 5.7] | 5.7 [5.2 to 6.2]
  Per protocol analyses: number analyzed (Participants) | 176 | 175
  Per protocol analyses | 5.5 [5.0 to 6.1] | 5.8 [5.3 to 6.3]
Statistical Analysis 1: Comparison: Intervention vs Control; Intent to treat population (all participants who were randomized, met pre-randomization eligibility criteria and who have post-enrollment follow-up data) was used for this analyses; Test type: Non-Inferiority — We estimated that we would need to enrol 700 women after taking into account the anticipated loss-to follow-up in order to provide 90% power to demonstrate whether gel use in women attending family planning (intervention) services is similar to, but no more than 20% lower than, gel use among women attending CAPRISA research clinics (control); Univariate Linear Mixed Models were used to analyze primary outcome; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.16 to 0.21] — The least square mean from the intervention arm was the minuend and the least square mean from the control arm was the subtrahend; The primary endpoint was compared using univariate linear mixed model with compound symmetry structure
Statistical Analysis 2: Comparison: Intervention vs Control; This is the analyses from the per protocol population (excluding all subsequent data collected from participants who were not dispensed product for more than 120 days); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Univariable Linear Mixed Models was used for the analyses; Median Difference (Final Values) = -0.25, 95% CI 2-sided [-0.98 to 0.48] — We calculated the difference in means between the two arms. The mean from the intervention arm was the minuend and the mean from the control arm was the subtrahend

2. Secondary Outcome: HIV Incidence Rates
Description: Time to HIV infection was calculated as the difference between estimated date of infection (midpoint between the last negative HIV test date and the first confirmed positive HIV test date) and enrolment date, plus one. Where a participant has a positive PCR and a negative rapid test on the same date, the date of infection is calculated as 14 days prior to this date. Women who do not become HIV positive before their last study visit will be censored on the day of their last negative HIV test. Their follow-up time will be calculated as the difference between date of censoring and enrolment date, plus one.
Time Frame: Between 2012 and 2015, up to 28 months
Population: Intent to treat population(all participants who were randomized, met pre-randomization eligibility criteria and who have post-enrollment follow-up data).
Measure: Number (95% Confidence Interval); unit: Incidence rate/100 women years
Groups:
- Intervention: 1% tenofovir gel provision through a public sector family planning services with 2-3 monthly provision and monitoring and the use of Quality Improvement methodology to promote reliable service delivery
  1% tenofovir gel: Participants will be randomized to receive 1% tenofovir gel through either:
  * Public sector family planning services with 2-3 monthly provision and monitoring of 1% tenofovir gel and the use of Quality Improvement methodology to promote reliable service delivery (intervention arm), or
  * The CAPRISA research clinics with monthly provision and monitoring of 1% tenofovir gel (control arm).
Arm/Group | Intervention | Control
Number analyzed (Participants) | 189 | 183
Incidence rate/100 women years | 3.5 [1.8 to 6.0] | 3.6 [1.9 to 6.3]
Statistical Analysis 1: Comparison: Intervention vs Control; The power was not calculated for all the secondary outcomes; Test type: Superiority; p = 0.928, z-test; We used z-test to compare incidence rates between the arms. We did not use log-rank test because we did not present survival curves; Incidence rate ratio = 0.96, 95% CI 2-sided [0.40 to 2.35] — We calculated incidence rate ratio, where the HIV incidence rate for the intervention arm represents the numerator and the HIV incidence rate for the control arm represents the denominator

3. Secondary Outcome: Pregnancy Incidence Rates
Description: Time to pregnancy, was as the difference between the estimated date of conception and the enrolment date, plus one. The date of conception was defined as 14 days after the last normal menstrual period or the estimated date of delivery minus 40 weeks if the first date of last normal menstrual period is not available or the midpoint between the date of the first positive pregnancy test and the date of the previous negative pregnancy test. The censoring time for a woman who did not become pregnant during the study equals the difference between the calculated censoring date and the enrolment date, plus one.
Time Frame: Between 2012 and 2015, up to 28 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Incidence rate/100 women years
Arm/Group | Intervention | Control
Number analyzed (Participants) | 189 | 183
Incidence rate/100 women years | 4.9 [2.8 to 7.9] | 5.1 [2.9 to 8.3]
Statistical Analysis 1: Comparison: Intervention vs Control; Power was not calculated for all the secondary outcomes; Test type: Superiority; p = 0.895, z-test; We used z-test to compare pregnancy incidence rates between the arms. We did not use log-rank test because we did not present survival curves; incidence rate ratio = 0.96, 95% CI 2-sided [0.45 to 2.04] — We calculated incidence rate ratio, where the pregnancy incidence rate for the intervention arm represents the numerator and the pregnancy incidence rate for the control arm represents the denominator

4. Secondary Outcome: Percentage of Participants Achieving Adherence >80%.
Description: Self-reported adherence to the tenofovir gel dosing strategy.Gel adherence was defined as the estimated proportion of reported sex acts covered by two gel doses and calculated for each woman by dividing half the number of returned used applicators each month by the number of reported sex acts that month.For participants attending 2-3 monthly clinic visits, their number of gels used in the last 30 days will be estimated as the total number of returned used gels, divided by the number of days between the current and the previous visit, times 30.
Time Frame: Between 2012 and 2015, up to 28 months
Population: This is a subset of intent to treat population. It includes all participants who returned used gel applicators and also reported sex during follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 188 | 181
percentage of participants | 70.2 [63.1 to 76.7] | 65.2 [57.8 to 72.1]
Statistical Analysis 1: Comparison: Intervention vs Control; Power was not calculated for all secondary outcomes; Test type: Superiority; p = 0.304, Regression, Log-binomial; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.94 to 1.24]

5. Secondary Outcome: HIV Viral Load Among HIV Seroconverters
Description: This is mean log transformed HIV viral load measured at the first visit post HIV infection.
Time Frame: Between 2012 and 2015, up to 28 months
Population: All participants who became HIV infected
Measure: Mean (Standard Deviation); unit: log10 copies/ml
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 12
log10 copies/ml | 4.4 (1.3) | 4.8 (0.9)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.455, t-test, 2 sided

6. Secondary Outcome: Tenofovir Resistance Among HIV Seroconverters
Time Frame: Between 2012 and 2015, up to 28 months
Population: Due to lack of funding, tenofovir resistance testing was not done in this study. However, we do have stored samples to fall back onto, should we secure funding.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Human Papillomavirus Incidence Rates
Description: For the calculation of the incidence rate, seroconversion was assumed to have occurred at the midpoint between the first positive HPV test and the previous HPV negative test.
Time Frame: Between 2012 and 2015, up to 28 months
Population: This is the subset of intent to treat population. It includes all participants who had HPV negative results at randomisation.
Measure: Number (95% Confidence Interval); unit: Incidence rate/100 women years
Arm/Group | Intervention | Control
Number analyzed (Participants) | 166 | 168
Incidence rate/100 women years | 1.0 [0.2 to 2.9] | 3.0 [1.4 to 5.8]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.097, z-test; incidence rate ratio = 0.33, 95% CI 2-sided [0.06 to 1.32] — We calculated incidence rate ratio, where the HPV incidence rate for the intervention arm represents the numerator and the HPV incidence rate for the control arm represents the denominator

8. Secondary Outcome: Percentage of Participants With Detectable Tenofovir Levels From Vaginal Samples at 12 Months of Follow-up
Description: Percentage of participants with detectable tenofovir levels from vaginal samples at 12 months of follow-up. All drug levels below limit of quantification were considered to be undetectable.
Time Frame: All participants with drug levels at 12 months of follow-up
Population: All participants with drug levels measured at 12 months of follow-up
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 157 | 156
percentage of participants | 39.5 [32.2 to 47.3] | 43.6 [36.1 to 51.4]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.462, Regression, Log-binomial; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.70 to 1.18]

9. Secondary Outcome: Product Acceptability
Description: This is the number of participants who reported that they liked the study product. The questionnaire was administered at study exit, therefore participants who were loss to follow-up and those who died could not complete the questionnaire.
Time Frame: At study completion, up to 28 months
Population: Participants who completed product acceptability questionnaire at study exit
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 184 | 177
Participants | 180 | 170

ADVERSE EVENTS:
Time Frame: Between 2012 and 2015, up to 28 months.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/189 | 2/183
Serious Adverse Events (participants affected / at risk) | 13/189 | 17/183
Other Adverse Events (participants affected / at risk) | 166/189 | 181/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=189) | Control (N=183)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal sphincter atony (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Investigation (Investigations) | 0 (0) | 1 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Anoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Caesarean section (Surgical and medical procedures) | 5 (5) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=189) | Control (N=183)
Conjunctivitis allergic (Eye disorders) | 4 (4) | 14 (14)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 17 (17)
Abdominal pain lower (Gastrointestinal disorders) | 14 (15) | 17 (19)
Diarrhoea (Gastrointestinal disorders) | 21 (22) | 45 (60)
Body tinea (Infections and infestations) | 13 (15) | 17 (18)
Gastroenteritis (Infections and infestations) | 11 (13) | 7 (7)
Influenza (Infections and infestations) | 15 (20) | 18 (22)
Nasopharyngitis (Infections and infestations) | 23 (27) | 66 (112)
Pelvic inflammatory disease (Infections and infestations) | 8 (9) | 16 (19)
Tonsillitis (Infections and infestations) | 20 (22) | 25 (31)
Upper respiratory tract infection (Infections and infestations) | 27 (36) | 24 (34)
Urinary tract infection (Infections and infestations) | 15 (15) | 17 (20)
Vaginitis bacterial (Infections and infestations) | 11 (12) | 14 (14)
Vulvovaginitis (Infections and infestations) | 25 (29) | 39 (49)
Blood pressure diastolic increased (Investigations) | 42 (50) | 27 (31)
Blood pressure increased (Investigations) | 22 (26) | 11 (13)
Blood pressure systolic increased (Investigations) | 42 (53) | 20 (27)
Abnormal loss of weight (Metabolism and nutrition disorders) | 11 (13) | 10 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 21 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 19 (19)
Headache (Nervous system disorders) | 28 (30) | 62 (91)
Genital ulceration (Reproductive system and breast disorders) | 10 (10) | 15 (16)
Vaginal discharge (Reproductive system and breast disorders) | 67 (91) | 73 (102)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 26 (33)
Hypertension (Vascular disorders) | 18 (18) | 11 (14)

LIMITATIONS AND CAVEATS:
The 2-3 monthly intervals between clinic appointments in the control arm is likely to introduce recall bias in this arm, unlike the monthly intervals in the intervention arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No